CLINICAL TRIAL: NCT02308332
Title: Effect of SwitChing AtriPla to Eviplera on Neurocognitive and Emotional Functioning, ESCAPE Study
Brief Title: Effect of SwitChing AtriPla to Eviplera on Neurocognitive and Emotional Functioning
Acronym: ESCAPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, J.E. Arends, Infectious Diseases Physician, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABR50959
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Neurocognitive Decline; HIV Associated Neurocognitive Disorder
MeSH Terms: interventions — Emtricitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): patients switching from Atripla to Eviplera
  Interventions: Drug: Eviplera
- Control (No Intervention): patients remaining on Atripla

INTERVENTIONS:
Drug: Eviplera — switch from Atripla to emtricitabine/rilpivirine/tenofovir (Eviplera)
  Other Names: emtricitabine/rilpivirine/tenofovir
  Arms: Intervention

SUMMARY:
This study will evaluate the effects of switching Atripla to Eviplera on neurocognition measured by neuropsychological testing and functional MRI

DETAILED DESCRIPTION:
Efavirenz, an antiretroviral drug used for the treatment of human immunodeficiency virus 1 (HIV-1) infections, is known for its neurological and psychiatric adverse events. Efavirenz is part of Atripla®, a single tablet regimen (STR), currently the most prescribed antiretroviral drug in the Netherlands. Recently, a new STR has become available, Eviplera® containing a successor of Efavirenz, named Rilpivirin. It has been shown in the phase-3 ECHO and THRIVE studies that Atripla as well as Eviplera have excellent and comparable antiretroviral efficacy in naive HIV-infected patients. Furthermore, data from these studies have shown that Eviplera was associated with fewer neurological and psychiatric adverse events than Atripla over 48 weeks. However, this was only patient reported adverse events, not neuropsychological evaluation. Furthermore, they were treatment naïve for HIV. Moreover, there might be a bias in these kind of switch studies due to the fact that those patients who switch will mostly regard their new combination better than the old one. Contrary, data on the long term impact of Efavirenz on neuropsychological performance and symptoms are conflicting.

Objective: This study aims to investigate the effect of switching from Atripla to Eviplera on neurocognitive performances (neurocognitive testing) and imaging (functional MRI scanning) in virologically suppressed HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Male, between 30 and 50 years
* HIV-1 RNA < 50 copies/mL on screening visit
* on Atripla continuously for ≥6 months preceding the screening visit
* Have a HIV genotype prior to starting cART with Atripla with no known resistance to any of the study agents at any time in the past including, but not limited to RT mutations K65R, K101E/P, E138G/K/Q/R, Y181C/I/V, M184V/I and H221Y
* Negative TPHA or VDRL < 12 months prior to the screening visit
* no signs of an acute or chronic hepatitis C infection within the past 12 months before screening as defined in the Dutch guideline (Arends et al. Neth J Med 2011)
* No subjective neurocognitive complaints in the preceding 12 months
* willingness to take Eviplera together with food according to the manufacturer's prescriptions.
* Estimated glomerular filtration rate ≥50 mL/min (Cockcroft-Gault formula) on last routine measurement during outpatient clinic
* able to understand and comply to study procedures and to provide written informed consent

Exclusion Criteria:

* Non-native Dutch speakers
* Proven major depression through psychiatric consultation within the past year or on anti-depressant drugs (SSRI or TCA)
* Active or known from medical history past CNS opportunistic infections
* History of proven neurologic disease (e.g. multiple sclerosis, brain tumor, cerebrovascular event, etc)
* Active psychiatric disorders classified according to the DMS V criteria
* History or evidence of alcohol or drug abuse defined according to DSM V criteria
* TSH within normal reference values on last routine measurement during outpatient clinic
* Contraindications for undergoing an MRI; a pacemaker or metallic devices/foreign bodies in situ, proven claustrophobia.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the neurocognitive performance as measured by neuropsychological test composite score after 12 weeks in stable HIV-infected patients switched from Atripla to Eviplera compared to a control group of patients on Atripla. | 12 weeks
  Patients will undergo a neuropsychological test battery where multiple standardized test will be undertaken to assess 7 different domains; Verbal Fluency, Executive Functioning, Speed of Information Processing, Learning, Memory, Attention/Working Memory, Motor skills. Raw scores can be calculated per domain and as a composite score. Differences in mean changes in composite score between baseline and end of study will be assessed with a paired T-test. A p-value <0.05 will be considered statistically significant. Within-arm changes will be assessed using Wilcoxon signed rank tests, and between-group comparisons will be evaluated with Wilcoxon rank sum tests. Multivariate analyses will be performed to analyse differences in the primary endpoints between the study groups.

SECONDARY OUTCOMES:
to assess the correlation between neurocognitive improvement (neuropsychological evaluation) and functional imaging (fMRI) after switching Atripla to Eviplera | 12 weeks
  The aim is to investigate if there is a correlation between improvement on neuropsychological test scores after 12 weeks of Eviplera therapy, and changes on fMRI after 12 weeks of Eviplera therapy. If there is a correlation, that means fMRI could be used to evaluate neurocognitive decline. Basically, we will asses if there is a correlation between ∆neuropsychological score and ∆fMRI-score. Because this is ordinal data, we will use a Spearman rank-order correlation to calculate a correlation-coefficient.
to evaluate correlation between neurocognitive performance and health related quality of life measured by SF-36 total score after switching from Atripla to Eviplera. | 12 weeks
  The aim is if an improvement in neuropsychological test scores after 12 weeks of Eviplera therapy is correlated with an improvement of quality of life. Basically, we will assess if there is a correlation between ∆neuropsychological score and ∆SF-36 total score. Because this is ordinal data, we will use a Spearman rank-order correlation to calculate a correlation-coefficient.
to assess the emotional functioning measured by HADS total score after switching Atripla to Eviplera by using a paired T-test to calculate differences in mean changes between baseline and end of study | 12 weeks
to assess USER-P (total scores) after switching Atripla to Eviplera | 12 weeks
to assess drug levels of Efavirenz (as a component of Atripla) and Rilpivirin (as a component of Eviplera) in relation to changes in neurocognitive performance and fMRI in both patient groups. | 12 weeks
  With this study, we want to investigate the effect of switching Efavirenz (as a component of Atripla) to Rilpivirine (as a component of Eviplera) on neurocognition. Our hypothesis is that neurocognition (as measured by neuropsychological testing scores) will improve when switching from Efavirenz (as a component of Atripla). If that is the case, hypothetically a lower or higher drug level of Efavirenz (as a component of Atripla) could have an effect on neurocognition (as measured by neuropsychological test scores). We will assess the correlation between drug level of Efavirenz or Rilpivirine and changes in neurocognitive function as measured by neuropsychological testing, and fMRI changes by regression analyses using drug levels as an independent variable and neuropsychological test scores as a dependent variable.
to evaluate the usefulness of PROMIS instruments in HIV research | 12 weeks
  In our study, we will use the PROMIS instruments Anxiety, Depression, Sleep disturbance and Satisfaction with social roles and activities. These are all short forms containing 8 questions or statements. Patients are asked to rate the questions from 1-5 into which extent they believe them to be true; 1 being not at all and 5 being very much. For each short form, a score will be calculated by adding the values of the response to each question. PROMIS provides a score conversion table where the score can be translated into a T-score. This rescales the patient's score into a standardized score with a mean of 50 and a standard deviation of 10. In order to provide these results, PROMIS uses a calibration sample containing data from over 21000 respondents. Differences in mean changes between baseline and end of study, as well as between the two study groups will be calculated using a paired T-test.

CONTACTS AND LOCATIONS:
Overall Officials: Joop Arends, MD PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Oomen PGA, Hakkers CS, Arends JE, van der Berk GEL, Pas P, Hoepelman AIM, van Welzen BJ, du Plessis S. Underlying Neural Mechanisms of Cognitive Improvement in Fronto-striatal Response Inhibition in People Living with HIV Switching Off Efavirenz: A Randomized Controlled BOLD fMRI Trial. Infect Dis Ther. 2024 May;13(5):1067-1082. doi: 10.1007/s40121-024-00966-7. Epub 2024 Apr 20. PMID 38642238